CLINICAL TRIAL: NCT05392777
Title: Utility of Residual Syntax Score to Predict Outcome After Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmad Samir, Principal investigator - Consultant, Cairo University
Other Study IDs: MS-2-221
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Myocardial Infarction
Keywords: Residual syntax score; STEMI; NSTEMI; Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Residual syntax score — residual syntax score will be calculated as the conventional syntax score from the web based tool, but subtract the score of the culprit lesion(s) that are fixed (stented) in the index procedure.

SUMMARY:
The aim of this study is to evaluate the utility of residual syntax score after PCI of the culprit vessel for patients with AMI (STEMI or NSTEMI) to predict 6-months clinical outcomes.

DETAILED DESCRIPTION:
A- Study Design: Prospective cross-sectional analytic study

B- Study Protocol: After attaining written informed consents from eligible STEMI/NSTEMI patients for participation in this observational study, data collection will be as follows: -

1. Targeted history taking emphasizing on:

   * Age of the patient, gender, and other risk-factors as hypertension, diabetes mellitus, smoking, substance abuse, dyslipidemia or family history of premature CAD.
   * Symptoms as chest pain and time of onset, previous CAD related symptoms, therapies or revascularization procedures.
   * Any relevant comorbid conditions.
   * Time delays labelled as patient related delay, door-to-first medical contact, any delays of transfer, door-to-needle or -to-wire crossing will be recorded.
2. Examination:

   Targeted physical examination of the patients with special emphasis on heart rate, blood pressure at presentation, Killip class (I-to-IV), signs suggestive of mechanical complications (new murmurs, pulmonary edema or cardiogenic shock).

   Patient weight and height will be collected to assess for overweight and/or obesity.
3. Standard 12-leads surface electrocardiogram (ECG):

   It will be obtained to as part of initial diagnosis, identify rhythm disturbances (heart block or any other arrythmias).

   Non-standard ECG (right or posterior leads positioning) would be ordered as appropriate.
4. Echocardiography:

   A rapid targeted bed-side study will be performed pre-cath as appropriate to assess LV-systolic function, regional wall motion abnormalities and any mechanical complication. Priority will be clearly for reperfusion, thus if the bed-side study would result in further delay, it will not be performed.

   All patients will have a formal and complete echo study before hospital discharge.
5. Laboratory data:

   Venous blood sample will be obtained from all patients for biochemistry analysis. Cardiac biomarkers, complete blood count, coagulation profile, liver and kidney function testing, lipid-profile, CRP and glycated hemoglobin (HbA1c).
6. Coronary angiography:

Coronary angiography and PCI is considered the gold-standard modality of revascularization for ST-segment Elevation myocardial infarction and is recommended within 24 hours for the majority patients presenting with NSTEMI.

Coronary angiography and PCI will be performed according to standard protocol. Culprit vessel, culprit lesion type and characteristics, initial and final TIMI flow, presence and number of non-culprit lesions will be collected and tabulated. Residual syntax score (rSS), as a surrogate for non-culprit atherosclerotic disease burden, will be equated as the conventional syntax score but subtracting the score of the culprit lesion(s) that have been passivated in the index procedure.

C- Follow-up Patients will be followed up for at least six-months to ensure compliance to medical therapy and life style interventions, and to report outcome measures accurately, including major adverse cardiac events (MACE), rehospitalization, target lesion revascularization, other unplanned revascularization and/or heart failure.

D- Data analysis By the end of the study period, the residual syntax score (rSS) will be used as a stratification tool to assess its correlation with outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

- Acute myocardial infarction (STEMI or NSTEMI)

Exclusion Criteria:

* Refusal to participate in the study.
* In case of NSTEMI, patients with unrecognizable culprit lesion will be excluded.
* Patients with previous coronary bypass surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Human participants of both genders, above the age of 18 years, with acute myocardial infarction (STEMI and NSTEMI) coming for primary or urgent PCI, who accept to participate to this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Composite of major adverse cardiovascular events (MACE). | 6 months
  Composite of MACE (defined as; CV death, non-fatal MI, non-fatal stroke)

SECONDARY OUTCOMES:
Rates of myocardial infarction | 6 months
Rates of cerebrovascular stroke | 6 months
  clinical and imaging proven cerebrovascular stroke
Rates of ischaemia-deriven unplanned revascularization | 6 months
  For new myocardial infarction or unstable angina
Rates of heart failure manifestations | 6 months
  Symptoms and signs consistent with heart failure diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Samir, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided